CLINICAL TRIAL: NCT04307979
Title: Impact of Bulletproof Coffee on Metabolism, Inflammation and Cognitive Function
Brief Title: Acute High Fat Bulletproof Coffee vs Black Coffee on Metabolism, Inflammation and Cognitive Function in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Bulletproof Coffee; H19-02684 (Other: UBC Clinical Research Ethics Board)
Record Dates: First submitted 2020-02-04; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Leukocytosis; Triglycerides; Cognitive Function; Inflammatory Response
Keywords: Triglycerides; Leukocyte; Monocyte; Neutrophil; Activation; High-fat
MeSH Terms: conditions — Leukocytosis

STUDY DESIGN:
Intervention Model Description: Randomized double-blind crossover design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulletproof Coffee (Experimental): A black coffee (bullet proof coffee keurig pod) with 29 grams of added fat (1 tablespoon bullet proof brain octane medium chain triglyceride oil, and 1 tablespoon bullet proof grass fed ghee) blended for 20 seconds with butter scent that is added to the lid.
  Interventions: Dietary Supplement: High-fat coffee; Dietary Supplement: Black coffee
- Black Coffee (Placebo Comparator): Black coffee that is blended for 20 seconds with butter scent added to the top of the lid.
  Interventions: Dietary Supplement: High-fat coffee; Dietary Supplement: Black coffee

INTERVENTIONS:
Dietary Supplement: High-fat coffee — A high fat coffee that consists of 29 grams of added fat from grass fed ghee, and MCT oil.
Dietary Supplement: Black coffee — A regular black coffee with no added caloric content.

SUMMARY:
This study will determine whether acute ingestion of a high fat "Bulletproof Coffee" will lead to changes in plasma triglycerides, immune cell function, as well as cognitive function when compared to a black coffee.

DETAILED DESCRIPTION:
In a randomized crossover design, participants will consume a single bulletproof coffee or a single black coffee separated by ~7 days. Each visit commences in the morning after an overnight fast of 10-12 hours, with no exercise the day prior, no coffee consumption the morning of testing, and completion of a food log for dietary duplication prior to visit 2. A fasting blood draw is obtained and cognitive function tests administered, along with questionnaires to assess gastrointestinal distress, arousal, and hunger/fullness before coffee consumption. Following this, one of the coffee beverages is consumed (randomized to each visit). Cognitive testing and questionnaires are completed at 60 minutes after finishing the coffee, another blood draw at 90 minutes, and then cognitive testing, questionnaires and a final blood draw 180 minutes after consuming the coffee. This procedure is repeated during their second experimental visit, in which they consume the remaining coffee based on their randomization.

ELIGIBILITY:
Inclusion Criteria:

* Must be over the age of 18
* Must drink between 1-4 cups of coffee per day (on average)
* Must be able to tolerate lactose and dairy products
* Have not been sick for the past 3 weeks (immune function)
* Non smoker
* Must be able to fast for 10-12 hours

Exclusion Criteria:

* If you are required to take corticosteroids (immune function)
* Cannot understand or speak English
* Individual has an auto-immune disease and requires medication
* Individual is following a ketogenic diet
* Individual has allergy or sensitivity to dairy, coffee or caffeine or coconut oil
* Individual has hypertension

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma triglycerides | Change over 3 hours following beverage consumption
  Circulating triglycerides measured in mmol/L

SECONDARY OUTCOMES:
Cognitive function | Change over 3 hours following beverage consumption
  Measures of cognitive function including Stroop test, digit substitution, and reaction time measured via computerized test battery.
Immune Cell Activation | Change over 3 hours following beverage consumption
  Assessment of activation markers on monocytes and neutrophils measured as median fluorescence intensity by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data used for publication will be shared in a raw data format. This will include participant ID, and all participant characteristics with no personally identifying information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent form will be available immediately upon study publication. The statistical analytical plan will be outlined in detail in the manuscript, however if more details are required, these will be provided. All information will be provided for 36 months following publication of results.
Access Criteria: IPD will be provided to credentialed research institutions/university labs. This data may be used for meta-analyses as well as direction for pilot work and future studies. Upon query, it will be determined whether the requesting party is eligible to view the data, both to maintain anonymity of the participants, and to ensure adequate, ethical and responsible use of IPD.